CLINICAL TRIAL: NCT06842849
Title: Impact of a Physical Exercise Program on the Physical, Podiatric and Mental Health of the Adult Population in a Rural Area
Brief Title: Impact of a Physical Exercise Program in a Rural Area
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, CARMEN GARCÍA GOMARIZ, Assistant Professor of Nursing, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESS_01
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Old Age; Debility
Keywords: old adults; exercise; accelerometry
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise T0 (Experimental): Carrying out an exercise program one year in progress
  Interventions: Other: Exercise program
- Exercise T1 (Experimental): Carrying out an exercise program without prior exercise
  Interventions: Other: Exercise program
- Control (No Intervention): Control

INTERVENTIONS:
Other: Exercise program — Multimodal and multicompetent exercise program 2 days a week for 60 minutes and 1 day of walking exercise for 60 minutes.
  Arms: Exercise T0; Exercise T1

SUMMARY:
With this work we want to assess whether there are differences in the amount of physical activity per week, measured by accelerometry in 3 groups of subjects, where one group (G1) has been carrying out a PA program called "Enguera Sé Saludable" for a year. another group (G2) newly introduced to the same exercise program, and a control group (G3) that does not carry out an exercise program but declared itself active.

DETAILED DESCRIPTION:
Active aging, according to the World Health Organization (WHO), involves making the most of everything that contributes to physical, mental and social well-being throughout life, thus promoting improved quality of life, functionality and longevity in the most advanced stages of life, seeking to minimize disability. To achieve active aging, older people must remain active in all aspects: physical, social and mental. For this reason, the WHO recommends that older adults engage in moderate to vigorous physical activity (MVPA) of 150 minutes a week The objetive, To assess whether there are differences in the amount of MVPA per week, measured by accelerometry in 3 groups of subjects, where one group (G1) had been carrying out a PA program called "Enguera Sé Saludable" for a year, another group (G2 ) newly inserted into the same exercise program, and a control group (G3) that did not carry out an exercise program but declared itself active.

Analytical quasi-experimental study, with 3 groups. A group (G1) over 59 years of age, of both sexes who have been doing PA since the year before the start of the study, within the "Enguera Be Healthy" Program in the municipality of Enguera. Another group (G2) of both sexes, newly enrolled in the same exercise program over 59 years of age. A control group (G3) of 59 years of both sexes who do not carry out the exercise program, inhabitants of Enguera and apparently active. The data analyzed was obtained from the placement of an Actigraph model GT3X BT accelerometer for a week and the collection of data from the various instruments such as the measurement of blood pressure and weight using the Tanita BC Scale. -545N, the Tinetti scale, the Time Up & Go test, the Monopodal Test, the SPPB test, the Sit to Stand Test, the Borg scale, the IPAQ questionnaire and the FHSQ questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 59 years of age.
* Patients who comply with accelerometer times for 7 days.
* Patients who correctly complete the accelerometer registration sheet.
* Patients who complete the informed consent

Exclusion Criteria:

* Patients who do not wear the accelerometer 600 minutes a day for at least 3 days on weekdays and 480 minutes for at least 1 day on the weekend.
* Patients who suffer from illness during data collection.
* Patients who do not wear the accelerometer for 7 days. Be in IPAQ category 1 (low level of AF).

Min Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MVPA | 1 year
  Mooderate to vigorous amount of activity. Assess the amount of moderate to vigorous exercise during accelerometry for one week.

SECONDARY OUTCOMES:
Up & Go | 1 year
  Evaluate basic mobility in older people and their probable gait and balance disorders. 1. Tell the elderly person to sit in the chair with their back supported by the backrest.
  2. Ask the person to get up from the chair, walk at a normal pace for a distance of 3 meters, have the person turns around, walks back to the chair and sits down again. 3. Measure the time the older person takes the test. Timing begins when the person He starts to get up from the chair and ends when he returns to the chair and sits down.
  4. Give a test try Normal: <10 seconds.
  * Mild mobility disability: 11-13 seconds.
  * High risk of falls: >13 seconds
Tinetti | 1 year
  Test that analyzes certain variables to evaluate gait and balance. The higher the score, the better the performance. The highest score of the gait subscale is 12, for balance 16. The sum of both scores for fall risk. The higher the score>the lower the risk <19 High risk of falls
SPBB | 1 YEAR
  Short Physical Performance Battery is an instrument that evaluates three aspects of mobility: balance, walking speed and strength of movement.
  limbs or lower extremities to get up from a chair. Supports the probable detection of outcomes adverse events such as mortality and institutionalization, as well as their association with disability.
Sit to Stand Test | 1 year
  Assesses the functional strength of the lower limbs, A chair was required on a flat surface and the subject was asked not to lean on his arms to get up and sit down, therefore, he was given a test opportunity with the instruction not to lean on. The patient is informed that the test consists of performing as many repetitions as possible of getting up and sitting down in a chair during a period of 60 seconds and that the time elapsed to the tenth repetition of getting up and sitting down will be timed at the same time. .
IPAQ | 1 year
  To estimate the level of mobility of older people. It includes seven questions that ask how often, for how long, and with what intensity the individual performed both moderate and vigorous activities during the past week, questions about time spent walking, and time spent sitting.
FHSQ | 1 year
  Specific to foot health, measuring quality of life based on foot pain, functional competence, footwear, and overall foot health. The first section consists of 13 questions measuring. The second section consists of 20 questions with Likert-type responses in 4 items. In the last section, the individual's sociodemographic information is collected. Regarding the interpretation of the results, given that the questionnaire does not provide a total score, the individual's responses must be entered into a computer application that will quantify a score from 0 to 100, with 0 being the worst state of health and 100 being the best.
Bood pressure | 1 year
  systolic and diastolic blood pressure measurement
Sex | o week , basaline
  Sex
BMC | 1 year
  Body mass index

CONTACTS AND LOCATIONS:
Overall Officials: CARMEN GARCÍA GOMARIZ, Principal Investigator — UNIVERSITAT DE VALÉNCIA DEPARTAMENTO D'INFERMERIA
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No